CLINICAL TRIAL: NCT01788319
Title: Micropulse Laser Trabeculoplasty (532nm) Versus Conventional Laser Trabeculoplasty (532nm) in Open Angle Glaucoma Patients
Brief Title: Micropulse Laser Trabeculoplasty (532nm) Versus Conventional Laser Trabeculoplasty (532nm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: S55194
Record Dates: First submitted 2013-02-01; First posted 2013-02-11 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2013-02

CONDITIONS: Open Angle Glaucoma
Keywords: laser trabeculoplasty; glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- lasertrabeculoplasty (Experimental)
  Interventions: Procedure: lasertrabeculoplasty

INTERVENTIONS:
Procedure: lasertrabeculoplasty
  Other Names: Conventional (532nm)

SUMMARY:
This study will investigate if micropulse laser trabeculoplasty (532nm) is as effecttive as or better than the conventional laser trabeculoplasty (532nm), it might be a new treatment strategy for glaucoma patients. It is done with a laser device that can also be used for many other ophthalmic applications, thus reducing the economic burden of treatment.

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years old
* willing to sign an informed consent and able to comply the requirements of the study
* having no other ocular diseases besides glaucoma

Exclusion Criteria:

* history of ocular trauma
* intraocular surgery (except for phaco)
* pigment dispersion and exfoliation glaucoma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
to compare the intraocular pressure reduction with the micropulse laser trabeculoplasty (532nm) versus the conventional laser trabeculoplasty (532nm) | one year of follow-up

SECONDARY OUTCOMES:
Secondary the complication rate between the two techniques will be compared | one year of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Vandewalle, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Department of Ophthalmology, UZLeuven, Leuven, Belgium